CLINICAL TRIAL: NCT04035096
Title: The Effectiveness of High-dose Intravenous Vitamin c With Very Low Carbohydrate Diet for Terminal Colon Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201901083MINB
Record Dates: First submitted 2019-07-22; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Colon Cancer Stage Iv
Keywords: high dose vitamin C; very low carbohydrate diet
MeSH Terms: conditions — Colonic Neoplasms | interventions — Ascorbic Acid; Methods; Control Groups

STUDY DESIGN:
Intervention Model Description: Clinical trial ( Pilot study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The high-dose vitamin C with very low carbohydrate diet group (Experimental): 1. Initiation of High dose IVC therapy: start with 25g IVC biweekly for one week; 50g IVC biweekly for one week; 75g biweekly for one week.
  2. Blood vitamin C level measurement: Confirm the plasma vitamin C level above 350 mg/dl by Arkray company PocketChem VC ( Kyoto, Japan) from the 75g/dose
  3. Once the target blood level is confirmed, the dose remains g biweekly for 12 weeks. If the target blood level is below 350mg/dl, the dose will titrate up to 100 g/dose or maximal dose of 1.5g/kg/dose to achieve the target level. The blood vitamin C level will be checked again and record. The final dose will be kept for 12 weeks.
  4. The Riordan IVC protocol (Taiwan)
  5. Maintenance dose: 75-100g every 2 week will be maintained for additional 12 weeks
  6. The infusion schedule change within 2 weeks is accepted with the fixed frequency per week or month
  7. VLCD intervention in the first 12 weeks
  Interventions: Drug: Ascorbic Acid
- The control group (Active Comparator): 1. Selection of control group: stage IV colon cancer patients match for sex, age and chemotherapy /target therapy drugs
  2. Usual care
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Ascorbic Acid — 1. Start with IVC (intravenous ascorbic acid) 25 g biweekly, 50 g biweekly, and 75 g biweekly. If the target blood level is below 350mg/dl, the dose will titrate up to 100 g/dose or maximal dose of 1.5g/kg/dose to achieve the target level.
  2. The final dose will be kept for 12 weeks.
  3. Maintenance dose: 75-100g every 2 week will be maintained for additional 12 weeks
  Other Names: VLCD (very low carbohydrate diet) intervention in the first 12 weeks
  Arms: The high-dose vitamin C with very low carbohydrate diet group
Other: Control group — 1. Selection of control group: stage IV colon cancer patients match for sex, age and chemotherapy /target therapy drugs
  2. Usual care
  Arms: The control group

SUMMARY:
The purpose is to evaluate the effectiveness of high dose intravenous vitamin C (IVC) therapy plus very low carbohydrate diet (VLCD) for stage IV colon cancer (with KRAS and BRAF mutation ) with or without chemotherapy.

DETAILED DESCRIPTION:
High dose IVC induces pro-oxidant effects, inhibits energy metabolism, acts as cytotoxic effect, and induces cancer cell apoptosis and necrosis. The recent advance in Warburg effect makes a new direction in high dose IVC therapy. The Warburg effect is the enhanced conversion of glucose to lactate observed in tumor cells, even in the presence of normal levels of oxygen. Converting glucose to lactate, rather than metabolizing it through oxidative phosphorylation in the mitochondria, is far less efficient as less ATP is generated per unit of glucose metabolized. Therefore, a high rate of glucose uptake is required to meet increased energy needs to support rapid tumor progression..

Vitamin C shares very similar structure with glucose. The high-dose IVC gets accessibility to glucose transporter, with competition to glucose. Having a reduced level of blood sugar seems to be a necessary parameter to increase IVC's anticancer effectiveness. VLCD with high dose IVC showed effectiveness in case series.

The investigator's project is a single-centered, clinical trial (pilot study) for stage IV colon cancer patients with or without chemotherapy. The experimental group will receive high dose vitamin C 75 or 100g (with blood vitamin C level > 350 mg/dl) in 1000 ml distilled water in 2-hour infusion, twice per week for 12 weeks. Then maintenance dose is 75-100 g once per 2 weeks for 12 weeks. Very low carbohydrate diet will be executed for the first 12 weeks. The control group will be matched for age, sex and chemotherapy and target therapy medication. The control group will receive usual care. The primary outcome will be the response rate by computerized tomography (CT) of the chest, abdomen and pelvis at 12 weeks and 24 weeks. The secondary outcome will be the improvement of tumor markers (CEA and Ca199).

This is the first clinical trial of IVC therapy with VLCD for stage IV colon cancer in Taiwan and in the world. This innovation will give us a primitive answer on the effectiveness of IVC therapy with VLCD for cancers. Vitamin C is a cheap and harmless therapy. The study result will open a door for alternative cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* stage IV colon cancer
* with KRAS and BRAF mutation

Exclusion Criteria:

* G-6-PD deficiency,
* metastatic kidney disease,
* obstructive uropathy,
* nephrotic syndrome,
* under other alternative medicine treatment or intravenous vitamin treatment,
* pregnant or lactating women,
* impaired renal function with a serum creatinine ≥ 132.6µmol/L(1.5 mg/dL)
* significant fluid retention(pleural effusion, ascites, lower leg edema),
* terminal heart failure,
* incapability to make decision,

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline by computerized tomography of Chest, abdomen and pelvis | 12 weeks
  all the participants will be evaluated by CT of the chest, abdomen and pelvis for possible response to treatment, using the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria at 12 weeks by the same radiologist, who is blind to the patients group.

SECONDARY OUTCOMES:
Number of participants with changes of tumor markers | 12 weeks
  CEA, and Ca 199

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Ying Chen, MD, MHSc, Principal Investigator — Department of Family Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 2 years after study completed.
Access Criteria: crystalcychen@ntu.edu.tw